CLINICAL TRIAL: NCT00556049
Title: Phase II, Single Arm Trial of Combination Sunitinib and Gemcitabine in Sarcomatoid and/or Poor-risk Patients With Metastatic Renal Cell Carcinoma
Brief Title: Combination Sunitinib and Gemcitabine in Sarcomatoid and/or Poor-risk Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry); Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Dror Michaelson, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-212
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Renal Cell Carcinoma; Neoplasm Metastases
Keywords: mRCC; sunitinib; gemcitabine
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Gemcitabine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sunitinib and gemcitabine
  Interventions: Drug: Gemcitabine; Drug: Sunitinib

INTERVENTIONS:
Drug: Gemcitabine — Intravenously on days 1 and 8 of each 21-day treatment cycle.
  Other Names: Gemzar
Drug: Sunitinib — Orally on days 1-14 of each 21-day treatment cycle
  Other Names: Sutent

SUMMARY:
The purpose of this research study is to determine if the combination of sunitinib and gemcitabine is effective in treating patients with metastatic renal cell carcinoma. The safety of this combination will also be studied. Sunitinib is approved by the FDA for the treatment of renal cell carcinoma. However, some patients' cancers do not respond to treatment or stops responding after initially responding. Gemcitabine is a chemotherapy drug that is approved by the FDA for the treatment of pancreatic cancer and several other cancers. It is not approved for the treatment of renal cell carcinoma. Previous research has suggested that combining gemcitabine with sunitinib may have some effectiveness in treating metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
* Participants will receive study treatment as an outpatient. Study treatment will be given in 3-week cycles.
* Sunitinib will be taken orally once per day for the first two weeks (days 1-14) of each treatment cycle.
* Gemcitabine will be given intravenously at the study clinic on days 1 and 8 of each treatment cycle.
* Before receiving sunitinib and gemcitabine on day 1 of each cycle the following will be performed: physical exam, performance status assessment and blood work. Before receiving gemcitabine on day 8 the following will be performed: physical exam, performance status assessment and blood work. Every 3 cycles a CT scan will be performed to measure the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic renal cell carcinoma with any sarcomatoid histology or poor-risk features as defined by having 3 or more of the following characteristics:

  * PS > 1, high serum lactate dehydrogenase
  * low hemoglobin
  * high "corrected" serum calcium
  * 2 or more sites of metastatic disease
  * time from initial diagnosis to evidence of metastatic disease 12 months or less
* Evidence of unidimensional measurable disease based on RECIST criteria, with at least 1 measurable lesion
* Male or female, 18 years of age or older
* ECOG performance status of 0-2
* Patients with brain metastasis can only be included of they were treated 4 weeks or more prior to enrollment with whole brain radiation and the effects of treatment have resolved
* Resolution of all acute toxic effects of prior therapy, radiotherapy or surgical procedure to NCI CTCAE version 3.0 grade of 1 or less
* Laboratory values as outlined in the protocol
* 2 weeks or more must have elapsed from the time of major surgery or radiation therapy prior to the day of registration
* No anticipated need for major surgical procedure during the course of the study

Exclusion Criteria:

* Prior treatment with sunitinib or gemcitabine
* More than one prior systemic therapy of any kind for renal cell carcinoma
* Uncontrolled high blood pressure
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack, or symptomatic congestive heart failure
* Ejection fraction < 30%
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* NCT CTCAE grade 3 or higher hemorrhage within 4 weeks of starting treatment
* Significant vascular disease
* Current grade 3 or higher cardiac dysrhythmia or QT prolongation
* Concurrent use of proarrhythmic medications including terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, and flecainide
* Pregnancy or breastfeeding or inadequate contraception
* Evidence of bleeding diathesis or coagulopathy
* Serious, non-healing wound, ulcer or bone fracture
* Psychiatric illness/social situation that would limit compliance with study requirements
* Previous diagnosis of concurrent malignancy requiring active systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Dror Michaelson, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center', Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Sunitinib and gemcitabine
  Gemcitabine: Intravenously on days 1 and 8 of each 21-day treatment cycle.
  Sunitinib: Orally on days 1-14 of each 21-day treatment cycle
Period: Overall Study
Arm/Group | Treatment
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 58 [45 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Overall Response Rate of Combination Therapy With Gemcitabine and Sunitinib in Sarcomatoid and/or Poor-risk mRCC Patients as First Line Therapy.
Time Frame: Until disease progression
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 72
percentage of participants | 25

ADVERSE EVENTS:
Groups:
- Neutropenia: Sunitinib and gemcitabine
  Gemcitabine: Intravenously on days 1 and 8 of each 21-day treatment cycle.
  Sunitinib: Orally on days 1-14 of each 21-day treatment cycle
Arm/Group | Neutropenia
Serious Adverse Events (participants affected / at risk) | 20/72
Other Adverse Events (participants affected / at risk) | 20/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neutropenia (N=72)
Neutropenia (Blood and lymphatic system disorders) | 20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neutropenia (N=72)
Neutropenia (Blood and lymphatic system disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No